CLINICAL TRIAL: NCT04158778
Title: Open-Label Proof of Concept Feasibility Study to Explore the Safety, Tolerability and Potential Role of MDMA-Assisted Psychotherapy for the Treatment of Detoxified Patients With Alcohol Use Disorder
Brief Title: Bristol Imperial MDMA in Alcoholism Study
Acronym: BIMA
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BIMA2016; 2016-002547-42 (EudraCT Number)
Record Dates: First submitted 2019-01-31; First posted 2019-11-12 (Actual); Last update posted 2019-11-12 (Actual); Status verified 2019-11

CONDITIONS: Alcohol Use Disorder
Keywords: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism | interventions — N-Methyl-3,4-methylenedioxyamphetamine; Psychotherapy

STUDY DESIGN:
Intervention Model Description: Open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- MDMA assisted Psychotherapy (Experimental): All participants receive 2 sessions of MDMA-assisted psychotherapy
  Interventions: Drug: MDMA; Other: Psychotherapy

INTERVENTIONS:
Drug: MDMA — Two sessions of MDMA-assisted psychotherapy will take place (session 3 & 7) within the 10 week course of psychotherapy. An initial dose of 125mg MDMA will be followed by an optional dose of 62.5mg 2 hours later.
  Other Names: 3,4-methylenedioxymethamphetamine
Other: Psychotherapy — Two sessions of MDMA-assisted psychotherapy will take place (session 3 & 7) within the 10 week course of psychotherapy.

SUMMARY:
The Safety, Tolerability and Role of MDMA-Assisted Psychotherapy for the treatment of detoxified patients with Alcohol Use Disorder.

DETAILED DESCRIPTION:
This is an open label within-subject feasibility study, in 20 patients with Alcohol Use Disorder who have recently undergone detoxification. All patients will receive MDMA-Assisted drug therapy. This study aims to assess if MDMA-Assisted Psychotherapy can be delivered safely and can be tolerated by patients with alcohol use disorder post-detoxification. Outcomes regarding abstinence from alcohol, quality of life and psychosocial functioning will be evaluated.

ELIGIBILITY:
Inclusion Criteria

* Informed consent
* Primary diagnosis (as defined by DSM-5) of alcohol use disorder.
* Successful alcohol detoxification (no longer consuming any alcoholic substances).
* Between 18 and 65 years old.
* Be able to identify in advance a supportive significant other(s):

  * who could accompany the patient to study visits if required -who can be contacted by the study team in order to remind the patient about follow- up appointments or collect outcome data (such as drinking behaviour) in the event that the patient themselves cannot be contacted.
* Proficient in speaking and reading English.
* Agree to comply with requirements of protocol.

Exclusion Criteria

* Lacking capacity
* History of, or a current, primary psychotic disorder, bipolar affective disorder type 1 or personality disorder;
* Present a serious suicide risk; this will be determined using the clinical judgement of the qualified mental health professionals within the research team. They will use information from the Columbia-Suicide Severity Risk Scale (C-SSRS) which allows classification of severity of suicidal ideation and behaviour. This scale classifies severe risk as a) current suicidal ideation with intent and/or plan; b) suicidal behaviour in the last 3 months. A clinical judgement regarding the level of risk and subsequent decisions regarding eligibility and care would use a combination of the information provided by the C-SSRS, the participant's history of previous risk behaviours, any presenting mental health difficulties and environmental and clinical factors. A final decision would usually include a discussion with qualified mental health professionals within the research team.
* Relevant abnormal clinical findings at screening visit judged by the investigator to render subject unsuitable for study. Including but not limited to:

  * History of cardiac disease, hypertension and stroke
  * History of severe liver disease, as evidenced by abnormal liver function test results, particularly reduction in albumin (normal > to 3.5 gm/dl).
  * History of epilepsy;
  * History of Malignant Hyperthermia (Central Core Disease);
* Regular user of Ecstasy (material represented as containing MDMA). E.g. more than five times in the last five years or at least twice in the 6 months prior to the start of the study;
* Currently taking or unwilling/unable to stop any medications inhibiting CYP 2D6, and the following medications Monoamine Oxidase Inhibitors, Ritonavir (HIV treatment), paroxetine, fluoxetine, citalopram, regular benzodiazepines or any other medications likely to interact with MDMA the opinion of the investigators, during 8 week MDMA assisted therapy only
* Regular use of/dependence on other drugs such as benzodiazepines, synthetic cannabinoids, cocaine and heroin.
* For females of childbearing age/potential

  * Must use an effective form of birth control for at least six days after administration of MDMA
  * Must not be pregnant and/or breast-feeding, until the end of the treatment phase.
* For males with partners of childbearing age/potential

  * Must themselves confirm use of an effective form of birth control for at least six days after administration of MDMA and confirm their partner will also, defined in detail in protocol.
* Taken part in a study involving an investigational product in the last three months
* Patients that might face additional risks from immunosuppression (for example patients with immunological diseases, patients with active infection or history of infections within 4 weeks of MDMA administration, etc).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-04-18 (Actual); Primary Completion 2020-06-12 (Estimated); Study Completion 2020-06-12 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability as measured by adverse event | Treatment period defined as: From first attendance for a psychotherapy session (Session 1) to the last psychotherapy session (session 10, approximately 8 weeks from treatment start).
  Number of patients completing 8-week course of MDMA-assisted psychotherapy.
  * Number of patients accepting second booster dose of MDMA during MDMA drug- assisted psychotherapy sessions.
  * All adverse events/reactions during the study will be tabulated, serious adverse events/ reactions will be coded according to CTCAE v4. The number of participants with treatment-related adverse events during the treatment period will be reported.

SECONDARY OUTCOMES:
Intensity of MDMA drug effect during MDMA-assisted psychotherapy sessions | MDMA-assisted psychotherapy sessions, at dosing and hourly for up to 8 hours after dosing.
  Intensity of drug effect assessed by verbal analogue scale 0 (none) 10 (most intense drug effect), participant and observer scores recorded.
Degree of psychological (subjective) distress (SUDS), participant and observer scores | MDMA-assisted psychotherapy sessions, -1 hour before dosing, at dosing and hourly following dosing for 8 hours. P
  Subjective Units of Distress scale (SUDS), degree of psychological (subjective) distress, rated from 0 (not at all distressed/completely relaxed) to 10 (most distressed imaginable/ panic attack). Participant and observer scores recorded.
Change in Vital signs during MDMA-assisted psychotherapy sessions: Heart Rate | MDMA-assisted psychotherapy sessions: 1 hour before dosing, at dosing, every 30 mins for 2 hours and hourly thereafter for 6 hours (extra measures taken if clinically required).
  The following will be measured 1 hour before dosing, at dosing, every 30 mins for 2 hours and hourly thereafter for 6 hours (extra measures taken if clinically required).
  -Heart rate (bpm) Pre-dosing measures will be compared to those taken after dosing.
Change in Vital signs during MDMA-assisted psychotherapy sessions: Temperature | MDMA-assisted psychotherapy sessions: 1 hour before dosing, at dosing, every 30 mins for 2 hours and hourly thereafter for 6 hours (extra measures taken if clinically required).
  The following will be measured 1 hour before dosing, at dosing, every 30 mins for 2 hours and hourly thereafter for 6 hours (extra measures taken if clinically required).
  -Temperature (degrees celsius) Pre-dosing measures will be compared to those taken after dosing.
Change in Vital signs during MDMA-assisted psychotherapy sessions: Systolic Blood pressure | MDMA-assisted psychotherapy sessions: 1 hour before dosing, at dosing, every 30 mins for 2 hours and hourly thereafter for 6 hours (extra measures taken if clinically required).
  The following will be measured 1 hour before dosing, at dosing, every 30 mins for 2 hours and hourly thereafter for 6 hours (extra measures taken if clinically required).
  Blood Pressure (mmHg) Pre-dosing measures will be compared to those taken after dosing.
Change in Vital signs during MDMA-assisted psychotherapy sessions: Diastolic Blood pressure | MDMA-assisted psychotherapy sessions: 1 hour before dosing, at dosing, every 30 mins for 2 hours and hourly thereafter for 6 hours (extra measures taken if clinically required).
  The following will be measured 1 hour before dosing, at dosing, every 30 mins for 2 hours and hourly thereafter for 6 hours (extra measures taken if clinically required).
  Blood Pressure (mmHg) Pre-dosing measures will be compared to those taken after dosing.
Subjective sleep following MDMA assisted psychotherapy | Daily for 7 days following both MDMA-assisted psychotherapy sessions (session 3 and 7).
  Leeds Evaluation Questionnaire, subjective, self-report measure, assessing changes in sleep quality and early morning behaviour. Visual analogue, positive end means improvement, negative ends mean decline in sleeping.
Mood rating during 7 days following MDMA assisted psychotherapy | Daily for 7 days following both MDMA-assisted psychotherapy sessions (session 3 and 7).
  Profile of Mood States questionnaire (POMS), a measure of mood states, 40 self-reported items, on a 5 point scale.
Acceptability of MDMA-Assisted therapy program: questionnaire | 2 months , completed at psychotherapy therapy sessions (1,2,3,4,5,6,7,8,9 & 10)
  Acceptability questionnaire designed for the study, this self report measure includes visual analogue scales and free text addressing the participants acceptability of taking part in the trial.
Change in Drinking behaviour | Baseline, Screening (day 0), Completed at psychotherapy therapy sessions, 1,2,3,4,5,6,7,8,9 & 10', Follow-up 3, 6, 9 months
  Drinking behaviour will be assessed using the clinician administered Time Line Follow Back scale- this tool allows collection of information about alcohol and illicit drug use. Pre-detoxification (screening visit) levels will be compared to levels at the final psychotherapy visit (session 10) and follow-up visits 3, 6 and 9 months. Any illicit drug use will also be recorded using this scale and assessed similarly.
Change in Quality of Life: SF-36 | Screening (day 0), 3, 6 and 9 months
  The Short Form Health Survey (SF-36). Gold standard, patient reported, quality of life questionnaire. Scores at follow-up visits, compared to screening/baseline.
Change in Subjective Sleep Quality: PSQI | Screening (day 0), 3, 6 and 9 months
  The Pittsburgh Sleep Quality Index. (PSQI). Sleep report questionnaire assessing the level of sleep disturbance. Scores collected at psychotherapy session 10 (final psychotherapy session), and follow-up visits compared to screening/ baseline.
Change in psychosocial functioning: Short Inventory of Problems for Alcohol (SIP) | Screening (day 0), 3, 6 and 9 months
  Short Inventory of Problems for Alcohol (SIP) Scale. This is a 15-item instrument assessing the self-attributable consequences of drinking. Scores collected at psychotherapy session 10 (final psychotherapy session), and follow-up visits compared to screening/ baseline.
Change in psychosocial functioning: Generalized Anxiety Disorder 7 (GAD-7) | Screening (day 0), 3, 6 and 9 months
  Generalized Anxiety Disorder 7 (GAD-7) scale. Brief self-administered questionnaire assessing anxiety. Scores collected at psychotherapy session 10 (final psychotherapy session), and follow-up visits compared to screening/ baseline.
Change in psychosocial functioning: The Patient Health Questionnaire (PHQ-9) | Screening (day 0), 3, 6 and 9 months
  The Patient Health Questionnaire (PHQ-9). Brief self-administered questionnaire assessing depressive symptoms.Scores collected at psychotherapy session 10 (final psychotherapy session), and follow-up visits compared to screening/ baseline.
Change in psychosocial functioning: Interpersonal reactivity Index (IRI) | Baseline, 3, 6 and 9 months
  Interpersonal reactivity Index (IRI) self-administered scale assessing aspects of empathy Scores collected at psychotherapy session 10 (final psychotherapy session), and follow-up visits compared to baseline.
Change in psychosocial functioning: The self compassion scale (SCS) | Baseline, psychotherapy session 10 (final psychotherapy session), follow-up visits at 3, 6 and 9 months
  The self compassion scale (SCS) self-administered scale assesses core aspects of self compassion including components of mindfulness. Scores collected at psychotherapy session 10 (final psychotherapy session), and follow-up visits compared to baseline.
The Penn Alcohol Craving Scale | Screening (day 0), 3, 6 and 9 months
  The Penn Alcohol Craving Scale (PACS) will assess craving, specifically frequency, intensity and duration of thoughts about drinking.Scores collected at psychotherapy session 10 (final psychotherapy session), and follow-up visits compared to baseline.
Obsessive Compulsive Drinking Scale | Screening (day 0), 3, 6 and 9 months
  Obsessive Compulsive Drinking Scale self-rated scale, used to measure obsessive and compulsive thoughts in relation to alcohol. Scores at psychotherapy session 10 (final psychotherapy session) and follow up visits will be compared to baseline
Prescribed medication use | Screening (day 0), 3, 6 and 9 months
  Prescribed medication use will be collected at every face-to-face visit and number and type of medications at psychotherapy session 10 (final psychotherapy session), and follow-up visits compared to screening/baseline.
Assessment of MDMA/Ecstasy use following MDMA-assisted therapy | Screening (day 0), session 10, 3, 6 and 9 months
  Participants will be asked to record any recreational MDMA use or craving to use recreational MDMA outside of the study.
Assessment of ability to collect follow-up data | Follow up 3,6 and 9 months
  Attrition at follow-up. Number of drop-outs at each visit.
Trauma History Questionnaire (THQ) | 2 month (Session 10)
  A self-report measure examining potentially traumatic experiences using a yes/no format. Administered on one occasion at the final therapy session (session 10)

CONTACTS AND LOCATIONS:
Overall Officials: Prof Nutt, Principal Investigator — Imperial College London
Locations (1):
- Study Center: University of Bristol, Bristol, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thurgur H, Sessa B, Higbed L, O'Brien S, Durant C, Wilson S, Szigeti B, Morgan CJA, Nutt DJ. MDMA-assisted psychotherapy for AUD: Bayesian analysis of WHO drinking risk level and exploratory analysis of drinking behavior and psychosocial functioning at 3 months follow-up. Alcohol Alcohol. 2025 May 14;60(4):agaf031. doi: 10.1093/alcalc/agaf031. PMID 40492610